CLINICAL TRIAL: NCT03984695
Title: Sexual Health Empowerment for Jail-Involved Women's Health Literacy and Prevention
Brief Title: Sexual Health Empowerment for Women's Health
Acronym: SHE-WOMEN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jason E Glenn, PhD, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00143316; 5R01CA181047-10 (NIH)
Record Dates: First submitted 2019-05-13; First posted 2019-06-13 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Breast Cancer; Contraceptive Usage; Sexually Transmitted Diseases
Keywords: Jail; Vulnerable Populations; STD Screening; unintended pregnancy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Breast Neoplasms; Contraception Behavior; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): * 15 minute discharge planning session with health educator
  * Health education booklet containing SHE-Women intervention content in print form(N~100)
  * access to health educator via text message
- Intervention (Experimental): Deliver text-Web intervention to (N ~100) women
  Researchers will deliver the integrated, multimedia electronic women's health literacy intervention arm of SHEWomen in text-Web format for individuals recently released from jail. Two health educators will be responsible for delivering content to participants, with an estimated contact time of ~10 hours pushed to participants over approximately a 5-day period.
  Interventions: Behavioral: SHE-WOMEN

INTERVENTIONS:
Behavioral: SHE-WOMEN — SHE-WOMEN is a text-Web intervention designed to increase jail-involved women's health literacy, reduce risk, and increase screening for prevention of cervical cancer, breast cancer, unintended pregnancy, and sexually transmitted infections.
  Arms: Intervention

SUMMARY:
The purpose of this study is to expand the reach of an existing cervical cancer literacy and prevention intervention- the Sexual Health Empowerment (SHE) Project . As a logical extension of the investigators earlier work, the objective of this renewal is to expand reach of SHE to address women's health disparities more broadly to create a sustainable model for dissemination of health promotion interventions for vulnerable populations.

DETAILED DESCRIPTION:
Over the last 35 years, there has been a 700% increase in the number of women in prisons and jails. These women, mostly women of color, have pervasive trauma histories, mental health problems, and drug use, all of which compromise their ability to engage in preventive health behaviors. For the last eight years, the research team has studied women leaving jail and why they are 4-5 times more likely to develop cervical cancer, a disparity that has remained unchanged for over 50 years. The original objective of the Sexual Health Empowerment (SHE) for Cervical Health Literacy and Prevention program (R01 CA181047) was to assess the effectiveness of a jail-based intervention to increase cervical health literacy and screening. SHE increased jailed women's cervical health literacy and rates of cancer screening after the women left jail.

While delivering SHE, researchers observed: 1) the cross-cutting nature of women's health risk factors, i.e. the risks that jailed women faced for cervical cancer also could lead to other women's health problems; and 2) opportunity for taking an evidence-based intervention, with a rich theoretical framing, to expand to other women's health issues faced by this group, around, not only cervical cancer prevention, but also breast cancer, unintended pregnancy, and STI prevention. While following women after release from jail (85% follow-up rate after 3 years), investigators also identified strategies for reaching this high-risk population through electronic communication. SHE participants were high users of mobile phones (88%), text (76%), Web (79%), and Facebook (70%). This renewal application presents an opportunity to holistically address health disparities experienced by women leaving jail and test new modalities for intervention delivery given use of electronic communication and social media.

The first aim uses an RCT to test the effectiveness of SHE-Women with women leaving jail on increasing women's health literacy, screening, and risk reduction practices (for cervical, breast cancer, unintended pregnancy, and STIs) against a standard of care. The second aim will be to understand the role and impact of human interaction in electronic interventions by tracking participants and interviewing key stakeholders.

Knowledge gained from this study will lead to an understanding of: 1) how a comprehensive women's health literacy intervention can narrow health disparities among justice-involved women and 2) the role of human interaction in successful electronic interventions, thereby creating a sustainable model for dissemination of health promotion interventions.

ELIGIBILITY:
Inclusion Criteria:

-Scheduled to leave jail within 3 days

Exclusion Criteria:

* not actively intoxicated
* not show severe psychological distress

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Glenn, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Jackson County Correctional Facility, Kansas City, Missouri, United States

REFERENCES:
- [Background] Ramaswamy M, Kelly PJ. "The Vagina is a Very Tricky Little Thing Down There": Cervical Health Literacy among Incarcerated Women. J Health Care Poor Underserved. 2015 Nov;26(4):1265-85. doi: 10.1353/hpu.2015.0130. PMID 26548678
- [Background] Ramaswamy M, Lee J, Wickliffe J, Allison M, Emerson A, Kelly PJ. Impact of a brief intervention on cervical health literacy: A waitlist control study with jailed women. Prev Med Rep. 2017 Apr 5;6:314-321. doi: 10.1016/j.pmedr.2017.04.003. eCollection 2017 Jun. PMID 28435785
- [Background] Nulsen FE, Becker DP. Control of hydrocephalus by valve-regulated shunt. J Neurosurg. 1967 Mar;26(3):362-74. doi: 10.3171/jns.1967.26.3.0362. No abstract available. PMID 6019745
- [Background] Guzman Silva MA. [Neuroendocrine cells (APUD) in adult human lung]. Acta Cient Venez. 1984;35(2):127-30. No abstract available. Spanish. PMID 6151327
- [Background] Stevens BJ. Mandatory continuing education for professional nurse relicensure. What are the issues? J Nurs Adm. 1973 Sep-Oct;3(5):25-8. No abstract available. PMID 4490746
- [Background] Steele RW, Hensen SA, Vincent MM, Fuccillo DA, Bellanti JA. A 51 Cr microassay technique for cell-mediated immunity to viruses. J Immunol. 1973 Jun;110(6):1502-10. No abstract available. PMID 4712922
- [Background] Sevilla CL, Fischer EH. The purification and properties of rat muscle glycogen phosphorylase. Biochemistry. 1969 May;8(5):2161-71. doi: 10.1021/bi00833a057. No abstract available. PMID 4306642
- [Background] Fernandez ME, Gonzales A, Tortolero-Luna G, Williams J, Saavedra-Embesi M, Chan W, Vernon SW. Effectiveness of Cultivando la Salud: a breast and cervical cancer screening promotion program for low-income Hispanic women. Am J Public Health. 2009 May;99(5):936-43. doi: 10.2105/AJPH.2008.136713. Epub 2009 Mar 19. PMID 19299678
- [Background] Guvenc G, Akyuz A, Acikel CH. Health Belief Model Scale for Cervical Cancer and Pap Smear Test: psychometric testing. J Adv Nurs. 2011 Feb;67(2):428-37. doi: 10.1111/j.1365-2648.2010.05450.x. Epub 2010 Oct 15. PMID 20946564
- [Background] Hogenmiller JR, Atwood JR, Lindsey AM, Johnson DR, Hertzog M, Scott JC Jr. Self-efficacy scale for Pap smear screening participation in sheltered women. Nurs Res. 2007 Nov-Dec;56(6):369-77. doi: 10.1097/01.NNR.0000299848.21935.8d. PMID 18004183
- [Background] Haynes MC, Ryan N, Saleh M, Winkel AF, Ades V. Contraceptive Knowledge Assessment: validity and reliability of a novel contraceptive research tool. Contraception. 2017 Feb;95(2):190-197. doi: 10.1016/j.contraception.2016.09.002. Epub 2016 Sep 9. PMID 27621043
- [Background] Melnick AL, Rdesinski RE, Creach ED, Choi D, Harvey SM. The influence of nurse home visits, including provision of 3 months of contraceptives and contraceptive counseling, on perceived barriers to contraceptive use and contraceptive use self-efficacy. Womens Health Issues. 2008 Nov-Dec;18(6):471-81. doi: 10.1016/j.whi.2008.07.011. Epub 2008 Oct 15. PMID 18926726
- [Background] Jaworski BC, Carey MP. Development and psychometric evaluation of a self-administered questionnaire to measure knowledge of sexually transmitted diseases. AIDS Behav. 2007 Jul;11(4):557-74. doi: 10.1007/s10461-006-9168-5. Epub 2006 Oct 3. PMID 17016760
- [Background] Helweg-Larsen M, Collins BE. The UCLA Multidimensional Condom Attitudes Scale: documenting the complex determinants of condom use in college students. Health Psychol. 1994 May;13(3):224-37. doi: 10.1037//0278-6133.13.3.224. PMID 8055858
- [Background] Brafford LJ, Beck KH. Development and validation of a condom self-efficacy scale for college students. J Am Coll Health. 1991 Mar;39(5):219-25. doi: 10.1080/07448481.1991.9936238. PMID 1783705

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: * 15 minute discharge planning session with health educator-This task was changed to a telephone session due to the COVID-19 Pandemic, which banned access to the recruitment sites.
  * Health education booklet containing SHE-Women intervention content in print form(N~100)
  * access to health educator via text message
- Intervention: Deliver text-Web intervention to (N ~100) women
  Researchers will deliver the integrated, multimedia electronic women's health literacy intervention arm of SHEWomen in text-Web format for individuals recently released from jail. Two health educators will be responsible for delivering content to participants, with an estimated contact time of ~10 hours pushed to participants over approximately a 5-day period.
  SHE-WOMEN: SHE-WOMEN is a text-Web intervention designed to increase jail-involved women's health literacy, reduce risk, and increase screening for prevention of cervical cancer, breast cancer, unintended pregnancy, and sexually transmitted infections.
- Pilot: These participants will give feedback on the digital, booklet, and survey items of the intervention
Period: Overall Study
Arm/Group | Control | Intervention | Pilot
Started | 127 | 128 | 24
Completed | 102 | 102 | 21
Not Completed | 25 | 26 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 127 | 128 | 255
Age, Continuous [Mean (Full Range); unit: years] | 39.83 [20 to 62] | 39.1 [23 to 67] | 39.45 [20 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 128 | 255
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Missing due to no response.
  Participants
    White: number analyzed (Participants) | 108 | 112 | 220
    White | 84 | 81 | 165
    Black: number analyzed (Participants) | 108 | 112 | 220
    Black | 9 | 9 | 18
    Hispanic: number analyzed (Participants) | 108 | 112 | 220
    Hispanic | 9 | 12 | 21
    Other: number analyzed (Participants) | 108 | 112 | 220
    Other | 6 | 10 | 16
Time Served in Jail or Prison (Lifetime) [Mean (Standard Deviation); unit: Months] — Population: Missing due to no response.
  Months
    Jail: number analyzed (Participants) | 126 | 125 | 251
    Jail | 21.33 (23.34) | 19.68 (28.20) | 20.49 (28.85)
    Prison: number analyzed (Participants) | 126 | 125 | 251
    Prison | 33.35 (47.63) | 30.95 (47.06) | 32.16 (47.23)

OUTCOME MEASURES:

1. Primary Outcome: Cervical Cancer Literacy
Description: Cervical Cancer Literacy Assessment Tool (C-CLAT) (PMID: 19299678) Adopted 16-items C-CLAT, the sum of scores on all 16 items reflects participants cervical cancer literacy with a possible total score ranges from 0 (minimum) to 16 (maximum).
  A higher score represents a higher level of cervical cancer literacy (i.e., better outcome).
Time Frame: Pre-Intervention assessment measured at baseline, Immediately post behavioral intervention assessment measured at 5 days after baseline, 12-month, 24-month, and 36-month follow-up assessments are measured accordingly after the baseline assessment
Population: There is missing data due to no response, measures reported are reported before multiple imputation for missingness (i.e., only complete cases).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 105 | 108
score on a scale
  Pre-Intervention assessment | 9.53 (2.95) | 9.05 (3.29)
  Post-intervention assessment: number analyzed (Participants) | 100 | 99
  Post-intervention assessment | 10.98 (2.67) | 11.51 (3.03)
  12-month assessment: number analyzed (Participants) | 75 | 75
  12-month assessment | 10.99 (2.41) | 11.07 (2.61)
  24-month assessment: number analyzed (Participants) | 61 | 53
  24-month assessment | 10.80 (2.09) | 11.38 (2.01)
  36-month assessment: number analyzed (Participants) | 24 | 19
  36-month assessment | 11.20 (2.12) | 11.21 (1.78)

2. Primary Outcome: Breast Cancer Literacy
Description: Breast Cancer Literacy Assessment Tool (B-CLAT) (PMID:23905580) Revised 22-items from B-CLAT (with an added item ask "At what age are most women supposed to start having mammograms?") The sum of scores on all 22 items reflects participants breast cancer literacy with a possible total score ranges from 0 (minimum) to 22 (maximum).
  A higher score represents a higher level of cervical cancer literacy (i.e., better outcome).
  ...items from revised Breast Cancer Literacy Assessment Tool (B-CLAT) (PMID:23905580) disagree or agree options: higher mean score = higher perception of risk
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 104 | 110
score on a scale
  Pre-Intervention assessment | 11.44 (3.99) | 10.92 (5.13)
  Post-Intervention assessment: number analyzed (Participants) | 100 | 98
  Post-Intervention assessment | 14.54 (3.75) | 15.45 (3.61)
  12-month assessment: number analyzed (Participants) | 75 | 75
  12-month assessment | 14.20 (3.48) | 15.04 (3.00)
  24-month assessment: number analyzed (Participants) | 61 | 53
  24-month assessment | 14.13 (2.84) | 14.53 (3.89)
  36-month assessment: number analyzed (Participants) | 24 | 19
  36-month assessment | 15.42 (2.62) | 14.84 (1.98)

3. Primary Outcome: Knowledge of Contraception
Description: -Contraceptive knowledge assessment (PMID:27621043) Adopted 8-items Contraceptive knowledge assessment, the sum of scores on all 8 items reflects participants cervical cancer literacy with a possible total score ranges from 0 (minimum) to 8 (maximum).
  A higher score represents a higher level of knowledge of contraception.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 103 | 104
score on a scale
  Pre-Intervention assessment | 5.33 (1.92) | 5.51 (1.96)
  Post-Intervention assessment: number analyzed (Participants) | 96 | 96
  Post-Intervention assessment | 6.53 (1.38) | 6.32 (1.68)
  12-month assessment: number analyzed (Participants) | 74 | 74
  12-month assessment | 6.55 (1.47) | 6.53 (1.55)
  24-month assessment: number analyzed (Participants) | 61 | 52
  24-month assessment | 6.59 (1.56) | 6.29 (1.74)
  36-month assessment: number analyzed (Participants) | 24 | 19
  36-month assessment | 6.88 (1.23) | 6.58 (1.26)

4. Primary Outcome: Beliefs About Acquisition and Use of Contraception
Description: -Beliefs about acquisition and use of contraceptive items from self-efficacy scale (PMID:18926726) Each item was on 5-point Likert scale range from 1 (Strongly Disagree) to 5 (Strongly Agree) A mean score of 10 items represent participants' beliefs of contraceptive barriers, ranges from 1 (minimum) to 5 (maximum).
  A higher score represents a higher level of perceived barriers (i.e., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 99 | 97
score on a scale
  Pre-Intervention assessment | 2.05 (0.75) | 2.05 (0.69)
  Post-Intervention assessment: number analyzed (Participants) | 96 | 96
  Post-Intervention assessment | 2.07 (0.82) | 1.94 (0.80)
  12-month assessment: number analyzed (Participants) | 74 | 73
  12-month assessment | 2.02 (0.75) | 1.92 (0.88)
  24-month assessment: number analyzed (Participants) | 60 | 53
  24-month assessment | 1.85 (0.81) | 1.88 (0.78)
  36-month assessment: number analyzed (Participants) | 24 | 19
  36-month assessment | 1.68 (0.55) | 1.93 (0.91)

5. Primary Outcome: Confidence in Use of Contraception
Description: -Beliefs about acquisition and use of contraceptive items from self-efficacy scale (PMID:18926726) Each item was on 5-point Likert scale range from 1 (Very confident) to 5 (Not at all confident).
  A mean score of reverse-coded 6 items represent participants' beliefs of contraceptive self-efficacy, ranges from 1 (minimum) to 5 (maximum).
  A higher score represents a higher level of contraceptive self-efficacy (i.e., better outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 96 | 96
score on a scale
  Pre-Intervention assessment | 2.92 (0.89) | 2.91 (0.96)
  Post-Intervention assessment: number analyzed (Participants) | 95 | 92
  Post-Intervention assessment | 3.13 (0.87) | 3.25 (0.77)
  12-month assessment: number analyzed (Participants) | 73 | 71
  12-month assessment | 3.08 (0.85) | 3.44 (0.68)
  24-month assessment: number analyzed (Participants) | 58 | 52
  24-month assessment | 3.26 (0.85) | 3.45 (0.73)
  36-month assessment: number analyzed (Participants) | 24 | 19
  36-month assessment | 3.24 (0.85) | 3.58 (0.48)

6. Primary Outcome: Knowledge of Sexually Transmitted Diseases
Description: -STD knowledge questionnaire (PMID: 17016760) Adopted 8-items STD knowledge questionnaire , the sum of scores on all 8 items reflects participants STD knowledge level with a possible total score ranges from 0 (minimum) to 8 (maximum).
  A higher score represents a higher level of knowledge of STD.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 95 | 96
score on a scale
  Pre-Intervention assessment | 4.28 (1.62) | 4.43 (1.63)
  Post-Intervention assessment | 5.24 (1.78) | 5.16 (1.33)
  12-month assessment: number analyzed (Participants) | 72 | 73
  12-month assessment | 4.82 (1.69) | 4.96 (1.46)
  24-month assessment: number analyzed (Participants) | 60 | 51
  24-month assessment | 4.67 (1.46) | 5.06 (1.69)
  36-month assessment: number analyzed (Participants) | 24 | 19
  36-month assessment | 5.46 (1.47) | 5.37 (1.61)

7. Primary Outcome: Confidence Using Condoms
Description: -Condom self-efficacy scale (PMID: 1783705) A mean score of 15 items were calculated with a possible range of 1 (minimum) to 7 (maximum).
  Higher scores represent a higher level of condom self-efficacy.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 100 | 99
score on a scale
  Pre-Intervention assessment | 4.24 (0.80) | 4.38 (0.72)
  Post-Intervention assessment: number analyzed (Participants) | 96 | 97
  Post-Intervention assessment | 4.35 (0.78) | 4.46 (0.69)
  12-month assessment: number analyzed (Participants) | 75 | 73
  12-month assessment | 4.45 (0.64) | 4.65 (0.53)
  24-month assessment: number analyzed (Participants) | 60 | 52
  24-month assessment | 4.53 (0.65) | 4.53 (0.65)
  36-month assessment: number analyzed (Participants) | 24 | 19
  36-month assessment | 4.64 (0.47) | 4.70 (0.38)

8. Primary Outcome: Attitudes Related to Condom Use
Description: -Multidimensional condom attitudes scale (PMID: 8055858) A mean score of 20-items was calculated with possible values range from 1 (minimum) to 7 (maximum).
  Items were rated on a 7-point scale ranging from strongly disagree to strongly agree.
  Higher mean score indicate more positive attitudes toward condoms.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 98 | 99
score on a scale
  Pre-Intervention assessment | 4.74 (0.84) | 4.77 (0.86)
  Post-Intervention assessment: number analyzed (Participants) | 97 | 97
  Post-Intervention assessment | 5.03 (0.84) | 5.08 (0.81)
  12-month assessment: number analyzed (Participants) | 75 | 74
  12-month assessment | 4.85 (0.72) | 5.09 (0.77)
  24-month assessment: number analyzed (Participants) | 59 | 52
  24-month assessment | 4.83 (0.89) | 5.13 (0.76)
  36-month assessment: number analyzed (Participants) | 24 | 19
  36-month assessment | 4.96 (0.59) | 5.21 (0.84)

9. Secondary Outcome: HPV Vaccination Receipt
Description: Behavioral Risk Factor Surveillance System (BRFSS) Human papillomavirus (HPV) vaccine question: have you ever had an HPV vaccination? A dichotomized score reflects participants' HPV vaccination receipt with 0 (no) and 1 (yes).
Time Frame: Only at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 89 | 87
Participants
  Not vaccinated | 70 | 62
  Vaccinated | 19 | 25

10. Secondary Outcome: Up to Date Pap Screening
Description: Health Information National Trends Survey-cervical cancer screening question: "When was your last pap screen?" A categorical items with four levels: 1) never; 2) within the past 3 years; 3) between 3 to 5 years; 4) 5 or more years ago.
Time Frame: Only at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 100 | 102
Participants
  Never | 1 | 2
  Within 3 years | 75 | 73
  3 to 5 years | 10 | 13
  Over 5 years | 14 | 14

11. Secondary Outcome: Up to Date Mammography
Description: Health Information National Trends Survey-breast cancer screening question: "When did you have your most recent mammogram to check for breast cancer? The items is only asked for participants over 50 years old. A categorical outcome with five levels: 1) never had a mammogram; 2) a year ago or less; 3) more than 1, up to 2 years ago; 4) more than 2 but no more than 5 years ago; 5) more than 5 years ago
Time Frame: Only at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 13 | 9
Participants
  Never | 1 | 1
  Less than a year | 2 | 5
  1 to 2 years | 4 | 1
  2 to 5 years | 5 | 2
  Over 5 years | 1 | 0

ADVERSE EVENTS:
Description: The behavioral intervention in the study includes access to online educational materials or a health education booklet, and there is no anticipated risk expected for participants, therefore the adverse event is not monitored.
Arm/Group | Control | Intervention | Pilot
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT03984695/Prot_SAP_000.pdf